CLINICAL TRIAL: NCT04299256
Title: Benson Relaxation Technique Combined With Music Therapy for Fatigue, Anxiety, and Depression in Hemodialysis Patients: A Randomized Controlled Study
Brief Title: Benson Relaxation Technique Combined With Music Therapy for Fatigue, Anxiety, and Depression in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Hacer Oturmaz, Clinical Nurse, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 4
Record Dates: First submitted 2020-03-05; First posted 2020-03-06 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Hemodialysis Complication; Fatigue; Anxiety Depression
Keywords: anxiety; depression; fatigue; hemodialysis; music therapy; relaxation
MeSH Terms: conditions — Fatigue; Anxiety Disorders; Depression | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Benson relaxation combined with music therapy (Experimental): In the first interview, the patient information delivered a training booklet explaining the definition, purpose, benefits and application techniques of BRT and music therapy to the patients in the intervention group. After patients reviewed the details in the training booklet, a weekly schedule was planned for each patient based on their hemodialysis days. For the initiation of the intervention, patients were invited to the hemodialysis unit at the hospital 45 min prior to their hemodialysis sessions. All the participants wore black eye patches to provide a dim environment and to focus better on their breath and the music piece. Then, the patients information opened the music piece and gave Benson Relaxation Technique comments in a slightly lower voice. Each session lasted for 20 min, and the music piece was switched off as Benson Relaxation Technique ended. The music piece used in the study was Daniel Kobelco's non-verbal classical song.
  Interventions: Behavioral: Benson relaxation combined with music therapy
- Control (No Intervention): Like the intervention group, the control group session (attention-matched education) which composed of 10-12 participants were performed with a booklet containing hemodialysis and its use in a silent room located in the hemodialysis units. The patient information provided in-person training on hemodialysis and its use for 20 min in a group session at the hemodialysis unit, on the first day of the study. During the study period, the participants in the control group were not subjected to any additional intervention.

INTERVENTIONS:
Behavioral: Benson relaxation combined with music therapy — In the first interview, the patient information delivered a training booklet explaining the definition, purpose, benefits and application techniques of BRT and music therapy to the patients in the intervention group. After patients reviewed the details in the training booklet, a weekly schedule was planned for each patient based on their hemodialysis days. For the initiation of the intervention, patients were invited to the hemodialysis unit at the hospital 45 min prior to their hemodialysis sessions. All the participants wore black eye patches to provide a dim environment and to focus better on their breath and the music piece. Then, the patients information opened the music piece and gave Benson Relaxation Technique comments in a slightly lower voice. Each session lasted for 20 min, and the music piece was switched off as Benson Relaxation Technique ended. The music piece used in the study was Daniel Kobelco's non-verbal classical song.
  Arms: Benson relaxation combined with music therapy

SUMMARY:
This study carried out in the HD unit of a large-scale training and research hospital, and at a dialysis center associated with this hospital located in Ankara, Turkey. Participants will be randomized to one of two study arms.

Arm 1: Intervention group Arm 2: Control group Hypothesis 1. The HD patients in the 8-week intervention of BRT combined with music therapy will report lower fatigue scores than those in the control group.

Hypothesis 2. The HD patients in the 8-week intervention of BRT combined with music therapy will perceive lower anxiety and depression than those in the control group.

DETAILED DESCRIPTION:
Patients undergoing hemodialysis treatment are susceptible to many complications. The inadequate stress-coping strategies render them vulnerable to high symptom burden and impaired quality of life. Patients are given conventional treatments to stop or slow down the progress of nephron destruction and prevent complications associated with uremia. However, previous studies observed that these therapies may be limited in alleviating fatigue, anxiety, and symptoms of depression, and may pose severe side effects. Therefore, in recent years patients have shown enhanced tendency to use complementary and integrative approaches including aromatherapy, acupuncture, massage, music, and relaxation to provide better control on their health and treatment process, feeling better physically, and emotionally, and as well as improve quality of life. The present study investigates the effects of Benson relaxation technique combined with music therapy in two-centered, 2-arm, assessor blinded randomized, controlled study of 61 hemodialysis patients.

Arm 1: Benson relaxation technique combined with music therapy ; Arm 2: control. The investigators hypothesize that Benson relaxation technique combined with music therapy will decrease severity of fatigue, anxiety, and depression.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were 18 years and older,
* Capable of communicating in Turkish,
* Had received HD in last three months,
* Undergone HD at least two times in a week,
* Showed a willingness to participate in this study.

Exclusion Criteria:

* Patients with aggravated conditions who would not be able to continue with the study,
* Other accompanying diseases that significantly affect the fatigue like COPD, advanced,
* Heart failure, asthma, and malignant tumors,
* Diagnosed with major depression,
* Could not communicate in Turkish,
* Used another complementary and integrative approach within the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Change in fatigue severity | Baseline measurements, at the end of 4th week, at the end of 8th week and two weeks after the completion of the interventions.
  Fatigue severity will be measured based on patient report by the Piper Fatigue Scale. Higher score means increase in fatigue severity.
Change in anxieyt and depression level. | Baseline measurements, at the end of 4th week, at the end of 8th week and two weeks after the completion of the interventions.
  Anxiety and depression will be measured by the Hospital Anxiety and Depression Scales. Higher scores on the scale mean worse anxiety and depression severity.

CONTACTS AND LOCATIONS:
Overall Officials: Hacer Oturmaz, MsC, RN, Principal Investigator — Hacettepe University
Locations (1):
- Ankara Training and Research Hospital Hemodialysis Units, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eroglu H, Gok Metin Z. Benson Relaxation Technique Combined With Music Therapy for Fatigue, Anxiety, and Depression in Hemodialysis Patients: A Randomized Controlled Trial. Holist Nurs Pract. 2022 May-Jun 01;36(3):139-148. doi: 10.1097/HNP.0000000000000509. PMID 35435875